CLINICAL TRIAL: NCT05493072
Title: Safety, Performance, and User Perceptions of RxConnect When Used to Provide Patient-specific, Indication Based Prescribing Support
Brief Title: RxConnect User Testing Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Imperial College London (Other)
Collaborators: National Institute for Health Research, United Kingdom (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 22CX7758
Record Dates: First submitted 2022-07-25; First posted 2022-08-09 (Actual); Results first posted 2025-03-24 (Actual); Last update posted 2025-03-24 (Actual); Status verified 2025-03

CONDITIONS: Behavior
Keywords: Medication safety; Prescribing practice; Prescribing behaviour
MeSH Terms: conditions — Behavior

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): Observation of control arm practice for 5 medication scenarios
- Intervention (Experimental): Observation of intervention practice for 5 medication scenarios
  Interventions: Other: RxConnect

INTERVENTIONS:
Other: RxConnect — Participants use RxConnect, an on-demand clinical decision support tool that receives medication and patient inputs and uses them to filter an underlying formulary, such as the BNF, and perform dosing calculations, as needed, to return patient-specific dosing recommendations.
  Arms: Intervention

SUMMARY:
Background

Medication errors are the leading cause of preventable harm in healthcare settings worldwide. An estimated 237 million medication errors occur in England alone every year, with 66 million considered clinically significant. There is an estimated cost to the NHS from definitely avoidable adverse drug reactions as a result of these errors of £98.5 million per year, consuming 181,626 bed-days and causing to 712 deaths.

Medication related clinical decision support systems, often integrated with electronic prescribing systems, are rapidly increasing in number over the last few decades, ranging from drug-drug interaction alerts to allergy checks and formulary support. A recent systematic review summarised that these systems are still relatively immature, with limited use of patient-specific input or human factors research used to develop them. There is an opportunity to improve these systems significantly for the benefit of the user and for patient safety. The World Health Organization propose that interventions to reduce medication error should include the development of technologies that are well understood and designed for the systems and practice they are applied to.

Human factors and usability engineering is an integral part of developing medical devices, such as clinical decision support (CDS) systems, to ensure that such devices are easy to use and can be used safely as intended. User testing / usability testing, which may incorporate several methods, should be conductive throughout the development process (at formative, summative assessment, and during post-market surveillance). These methods are now becoming more common place in healthcare technology research and should continue to support the development of new technologies.

RxConnect

RxConnect, a newly registered UKCA marked medical device, is an on-demand clinical decision support tool that receives medication and patient inputs and uses them to filter an underlying formulary, such as the BNF, and perform dosing calculations, as needed, to return patient-specific dosing recommendations. RxConnect does not have a user interface and relies on an integration with third-party systems, such as electronic prescribing systems, to deliver CDS services to clinical end users. For this study a prototype user interface for RxConnect that emulates a typical electronic prescribing system will be used.

The study team hypothesise that use of RxConnect as a digital prescribing aid is quicker, easier, and as safe to use as currently available prescribing aids. This study aims to utilise user testing to prove or disprove the above hypothesis and to generate quantitative and qualitative outputs to support the continued development of RxConnect prior to clinical deployment.

ELIGIBILITY:
Inclusion Criteria:

* Willingness to consent and participate
* Medical doctor - Foundation year 1 and above OR registered non-medical prescriber (e.g. nurses or pharmacists)
* Regular (at least weekly) experience in prescribing medications as part of working role

Exclusion Criteria:

* Infrequent prescribing practice (less than once a week)
* Not willing to participate

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2022-12-12 (Actual); Primary Completion 2023-03-30 (Actual); Study Completion 2023-03-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Imperial College NHS Healthcare Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Donaldson LJ, Kelley ET, Dhingra-Kumar N, Kieny MP, Sheikh A. Medication Without Harm: WHO's Third Global Patient Safety Challenge. Lancet. 2017 Apr 29;389(10080):1680-1681. doi: 10.1016/S0140-6736(17)31047-4. No abstract available. PMID 28463129
- [Background] MHRA. Guidance on applying human factors and usability engineering of medical devices including drug-device combination products in Great Britain. 2021;(January):35. Available from: https://assets.publishing.service.gov.uk/government/uploads/system/uploads/attachment_data/file/970563/Human-Factors_Medical-Devices_v2.0.pdf
- [Background] Holden RJ, Abebe E, Russ-Jara AL, Chui MA. Human factors and ergonomics methods for pharmacy research and clinical practice. Res Social Adm Pharm. 2021 Dec;17(12):2019-2027. doi: 10.1016/j.sapharm.2021.04.024. Epub 2021 May 2. PMID 33985892
- [Background] Novak LL, Holden RJ, Anders SH, Hong JY, Karsh BT. Using a sociotechnical framework to understand adaptations in health IT implementation. Int J Med Inform. 2013 Dec;82(12):e331-44. doi: 10.1016/j.ijmedinf.2013.01.009. Epub 2013 Apr 3. PMID 23562140
- [Result] Elliott RA, Camacho E, Jankovic D, Sculpher MJ, Faria R. Economic analysis of the prevalence and clinical and economic burden of medication error in England. BMJ Qual Saf. 2021 Feb;30(2):96-105. doi: 10.1136/bmjqs-2019-010206. Epub 2020 Jun 11. PMID 32527980
- [Result] Tolley CL, Slight SP, Husband AK, Watson N, Bates DW. Improving medication-related clinical decision support. Am J Health Syst Pharm. 2018 Feb 15;75(4):239-246. doi: 10.2146/ajhp160830. PMID 29436470
- [Result] Aufegger L, Serou N, Chen S, Franklin BD. Evaluating users' experiences of electronic prescribing systems in relation to patient safety: a mixed methods study. BMC Med Inform Decis Mak. 2020 Apr 3;20(1):62. doi: 10.1186/s12911-020-1080-9. PMID 32245467
- [Derived] Feather C, Clarke J, Appelbaum N, Darzi A, Franklin BD. Comparing safety, performance and user perceptions of a patient-specific indication-based prescribing tool with current practice: a mixed methods randomised user testing study. BMJ Qual Saf. 2025 Oct 17;34(11):737-746. doi: 10.1136/bmjqs-2024-017733. PMID 39577867

RESULTS

PARTICIPANT FLOW:
Groups:
- 1 - Control First, Then Intervention: Observation of control arm practice for 5 medication scenarios (using standard prescribing practice), then intervention arm for 5 medication scenarios (using the intevention to support prescribing practice).
- 2- Intervention First, Then Control: Observation of intervention arm for 5 medication scenarios (using the intevention to support prescribing practice).
  Then Observation of control arm practice for 5 medication scenarios (using standard prescribing practice)
Period: Overall Study
Arm/Group | 1 - Control First, Then Intervention | 2- Intervention First, Then Control
Started | 12 | 12
Completed | 12 | 12
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Study Participants: All study participants exposed to both control and intervention, therefore reported together
Arm/Group | All Study Participants
Number analyzed (Participants) | 24
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 24
  >=65 years | 0
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Gender: Female | 15
  Gender: Male | 8
  Gender: Not stated | 1
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Profession [Count of Participants; unit: Participants]
  Doctor | 20
  Pharmacist | 4
Speciality [Count of Participants; unit: Participants]
  Paediatric Emergency | 1
  Paediatric Intensive Care Unit | 4
  Paediatrics | 9
  Adults | 10
Participant grade (self reported titles used) [Count of Participants; unit: Participants]
  Foundation Year 1 | 1
  Senior House Officer | 1
  CT/ST Years 1-5 | 5
  ST Years 6-8 | 6
  Registrar | 1
  Clinical Fellow | 3
  Trust Grade | 2
  Consultant | 1
  Pharmacist Pay Band 8A | 1
  Pharmacist Pay Band 8B | 3
Years using Cerner [Count of Participants; unit: Participants]
  <1 year | 6
  1-2 years | 2
  2-3 years | 6
  3-4 years | 2
  4-5 years | 2
  5+ years | 6

OUTCOME MEASURES:

1. Primary Outcome: Number of Prescribing Errors by Study Arm
Description: Sub analysis of errors by type available in full report
Time Frame: 60 minutes
Measure: Count of Units; unit: Medication orders
Units Other Than Participants: Medication orders
Groups:
- RxConnect (Experiment Arm): Participants were asked to complete 5 test scenarios using Touchdose to determine the required dose recommendation. Participants were asked to 'trust' Touchdose and were reminded that they were not required to check or confirm the dose recommendations with any other resources or calculators. Participants entered the dose recommendation for each medication scenario for the required test patient on the Cerner Millennium Power Chart currently used at the study site for electronic prescribing.
- Current Practice (Control) Arm: Participants were asked to complete 5 test scenarios using the usual resources available to them in their prescribing practice. Access was provided to the prescribers usual electronic prescribing platform, including links to the British National Formulary, MedicinesComplete, local antimicrobial stewardship application, local intranet, and a generic online search engine. A hard copy of the BNF and BNFc was also readily available. Participants entered the dose recommendation for each medication scenario for the required test patient on the Cerner Millennium Power Chart currently used at the study site for electronic prescribing.
Arm/Group | RxConnect (Experiment Arm) | Current Practice (Control) Arm
Number analyzed (Participants) | 24 | 24
Number analyzed (Medication orders) | 120 | 120
Medication orders
  Erroneous medication order | 8 | 34
  Dose error | 8 | 31
  Route error | 3 | 4
  Patient error | 0 | 1
  Frequency error | 0 | 3
  Formulation error | 3 | 6

2. Secondary Outcome: Number of Medication Orders With a Large Magnitude Error (Greater Than 25% of the Recommended Dosing Range)
Description: Dosing errors with a deviation of more than 25% from the recommended range were categorised as large magnitude errors.
Time Frame: 60 minutes
Measure: Count of Units; unit: Medication orders
Units Other Than Participants: Medication orders
Arm/Group | RxConnect (Experiment Arm) | Current Practice (Control) Arm
Number analyzed (Participants) | 24 | 24
Number analyzed (Medication orders) | 120 | 120
Medication orders | 6 | 22

3. Secondary Outcome: Time Taken to Prescribe Each Medication
Description: For the first scenario, TTP was calculated from the moment the participant began reading the scenario to task completion, while for subsequent scenarios, timing started from the completion of the previous scenario. The endpoint for each scenario was marked by the participant's submission of the medication order on the electronic prescribing (eP) system.
Time Frame: 60 minutes
Measure: Mean (95% Confidence Interval); unit: seconds
Units Other Than Participants: Medication orders
Arm/Group | RxConnect (Experiment Arm) | Current Practice (Control) Arm
Number analyzed (Participants) | 22 | 22
Number analyzed (Medication orders) | 110 | 110
seconds | 179.7 [166.1831 to 193.2897] | 224.8 [205.2554 to 244.3992]

4. Secondary Outcome: Measurement of the Prescribers Perceived Mental Load Per Prescribing Scenario
Description: Measurement of the Prescribers perceived mental load per prescribing scenario, Using NASA task load index (TLX).
  An overall workload score combining all 6 NASA TLX domains was calculated (minimum 0 lower workload - maximum 126 highest workload).
Time Frame: 60 minutes
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | RxConnect (Experiment Arm) | Current Practice (Control) Arm
Number analyzed (Participants) | 24 | 24
score on a scale | 41.45 [33.02 to 49.89] | 57.21 [48.69 to 65.72]

5. Other Pre Specified Outcome: Erroneous Medication Orders by Hierarchial Task Analysis (Identifying Vulnerable Steps in the Prescribing Workflow).
Description: Erroneous orders identified as a primary outcome of the study will then be analysed using hierarchical task analysis (HTA). The HTA is a qualitative outcome, different from the primary outcome (error yes/no) by instead identifying 'where' within the prescribing process an error occurred.
  Workflow steps, representing tasks or actions in both the control and intervention arms, were developed based on established and anticipated prescribing workflows and refined as new, unanticipated steps emerged during study observations. These workflows were then employed for hierarchical task analysis, as detailed in the data analysis section.
  Hierarchical task analysis was conducted by reviewing recordings of all erroneous medication orders, breaking down the prescribing process into discrete steps. This structured approach allowed for identification of potential risks or inefficiencies in the workflow, helping trace each error's likely origin within the process.
Time Frame: 60 minutes
Measure: Number; unit: Medication orders
Units Other Than Participants: Medication orders
Arm/Group | RxConnect (Experiment Arm) | Current Practice (Control) Arm
Number analyzed (Participants) | 24 | 24
Number analyzed (Medication orders) | 120 | 120
Medication orders
  Overall erroneous medication orders | 8 | 34
  Review written patient scenario | 5 | 8
  Access prefered/necesary dosing resource | 0 | 1
  Identify medication, appropriate indication and dose recommendation | 0 | 7
  Identify any relevant dose considerations | 0 | 12
  Calculate dose as per resource directions | 0 | 3
  Condsider if any min/max dose constraints need taking into account | 0 | 1
  Select/search for or confirm route from unfiltered list | 0 | 1
  Select/search for form from unfiltered list | 0 | 1
  Launch required patient in Cerner | 1 | 0
  Select one or more dose recommendation(s) | 1 | 0
  Enter/confirm dose | 1 | 0

6. Other Pre Specified Outcome: Number of Participants That Gave Qualitative Feedback
Description: Audio of interviews will be transcribed verbatim and thematically analyses to provide insights from participants that can be utilised for recommendations for practice and research.
Time Frame: 60 minutes
Population: There is only one arm reported for the qualitative feedback as all participants provided feedback.
Measure: Number; unit: participants
Groups:
- Number of Participants That Gave Qualitative Feedback: All participants provided qualitative feedback as described in the Full study report
Arm/Group | Number of Participants That Gave Qualitative Feedback
Number analyzed (Participants) | 24
participants | 24

ADVERSE EVENTS:
Time Frame: 60 minutes
Groups:
- Current Practice (Control Arm): Participants exposed to both arms but in alternate orders.
  Participants were asked to complete 5 test scenarios using the usual resources available to them in their prescribing practice. Access was provided to the prescribers usual electronic prescribing platform, including links to the British National Formulary, MedicinesComplete, local antimicrobial stewardship application, local intranet, and a generic online search engine. A hard copy of the BNF and BNFc was also readily available. Participants entered the dose recommendation for each medication scenario for the required test patient on the Cerner Millennium Power Chart currently used at the study site for electronic prescribing.
- RxConnect (Experiment Arm): Participants exposed to both arms but in alternate orders.
  Participants were asked to complete 5 test scenarios using Touchdose to determine the required dose recommendation. Participants were asked to 'trust' Touchdose and were reminded that they were not required to check or confirm the dose recommendations with any other resources or calculators. Participants entered the dose recommendation for each medication scenario for the required test patient on the Cerner Millennium Power Chart currently used at the study site for electronic prescribing.
Arm/Group | Current Practice (Control Arm) | RxConnect (Experiment Arm)
All-Cause Mortality (participants affected / at risk) | 0/24 | 0/24
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/24
Other Adverse Events (participants affected / at risk) | 0/24 | 0/24

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-06-15): https://cdn.clinicaltrials.gov/large-docs/72/NCT05493072/Prot_SAP_000.pdf